CLINICAL TRIAL: NCT01883271
Title: Effect of Aerobic Interval vs. Continuous Exercise Training on Cardiovascular Function in Aging
Brief Title: Effect of Aerobic Interval Training on Cardiovascular Function in Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB201700044; 551-2012 (Other: University of Florida)
Record Dates: First submitted 2013-06-13; First posted 2013-06-21 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- High intensity aerobic interval training (Experimental): Older adults will complete 8 weeks of high intensity aerobic interval exercise training.
  Interventions: Other: High intensity aerobic interval training
- Continuous moderate intensity exercise (Experimental): Older adults will complete 8 weeks of continuous moderate intensity exercise training.
  Interventions: Other: Continuous moderate intensity exercise
- Non-exercise control group (No Intervention): Older adults assigned to the non-exercise control group will maintain their normal lifestyle for 8 weeks.
- Young Healthy controls (No Intervention): Young healthy subjects will be assigned to the healthy control group and will undergo baseline measures only.

INTERVENTIONS:
Other: High intensity aerobic interval training — Supervised aerobic interval training will be performed on bicycles 4 times per week for 8 weeks. Each training session will last 40 minutes and will consist of 10-minute warm up at 70% of maximal heart rate (HRmax), four 4-minute intervals at 90% of HRmax with 3-min active recovery at 70% of HRmax and 5-minute cool down at 70% of HRmax.
  Arms: High intensity aerobic interval training
Other: Continuous moderate intensity exercise — Supervised exercise training will be performed on bicycles 4 times per week for 8 weeks. Each training session will last 47 minutes and will consist of continuous moderate intensity cycling at 70% of HRmax.
  Arms: Continuous moderate intensity exercise

SUMMARY:
Study objectives:

1. To compare cardiovascular function in older compared to young healthy adults.
2. To compare the effect of 8 weeks of aerobic interval training vs. continuous moderate exercise on cardiovascular function in healthy older adults.

Hypotheses:

1. Compared to young adults, older adults will have lower cardiovascular function.
2. Compared to continuous moderate intensity exercise training, interval training will be more effective in improving cardiovascular function in older adults.

DETAILED DESCRIPTION:
Cardiovascular function will be measured at baseline in older healthy adults and young healthy controls. Older adults will be randomized to the aerobic interval training group, continuous moderate exercise group or non-exercise control group. At the end of the 8-week exercise intervention, baseline measures will be repeated in the older adults.

ELIGIBILITY:
Inclusion Criteria for older adults:

* Healthy men and women 55 to 79 years of age
* Sedentary or minimally physically active for at least the prior 1 year.
* Women will be premenopausal or postmenopausal (either natural or surgical) defined as a cessation of menses for at least 2 years.
* Premenopausal women will be eumenorrheic and will be studied during the early follicular phase (days 1 through 6) of the menstrual cycle.
* Able to give consent.

Inclusion Criteria for young adults:

* Healthy men and women 18 to 35 years of age
* Sedentary or minimally physically active for at least the prior 1 year.
* Women will be premenopausal, eumenorrheic and will be studied during the early follicular phase (days 1 through 6) of the menstrual cycle.
* Able to give consent.

Exclusion Criteria:

* history of diabetes
* history of any relevant cardiovascular diseases (myocardial infarction, angina pectoris, history of coronary artery bypass surgery or angioplasty, congestive heart failure, or arrhythmia)
* hypertension (≥160 mmHg systolic or ≥100 mmHg diastolic)
* history of renal impairment
* history of gout or hyperuricemia
* history of hepatic disease or infection with hepatitis B, C
* history of seizures, or other relevant on-going or recurrent illness
* recent (within 3 months) or recurrent hospitalizations
* use of tobacco products
* >5 % weight change in the prior 6 months.
* current intake of medications that may affect study results
* participation in regular aerobic exercise training (>30 minutes,

  * 3 times/wk in the past year).
* premenopausal women taking oral contraceptives and postmenopausal women taking hormone replacement therapy.
* pregnancy (positive urine pregnancy test) or lactation

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2019-02-21 (Actual); Study Completion 2019-02-21 (Actual)

PRIMARY OUTCOMES:
Change in vascular endothelial function | At baseline and after 8 weeks of exercise training
  Brachial flow-mediated dilation using ultrasonography

SECONDARY OUTCOMES:
Change in factors related with endothelial function | At baseline and after 8 weeks of exercise training
  Blood and cellular markers of oxidative stress and inflammation
Change in arterial stiffness | At baseline and after 8 weeks of exercise training
  Arterial stiffness and wave reflection will be measured using the SphygmoCor device
Change in cardiac function | At baseline and after 8 weeks of exercise training
  Left ventricular systolic and diastolic function will be measured using echocardiography
Change in maximal oxygen consumption | At baseline and after 8 weeks of exercise training
  Maximal oxygen consumption will be measured using online computer-assisted open-circuit spirometry during incremental treadmill exercise

CONTACTS AND LOCATIONS:
Overall Officials: Demetra D Christou, Ph.D, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States